CLINICAL TRIAL: NCT04688515
Title: Effectiveness of a Nutrition Program Using Positive Deviance Approach to Reduce Undernutrition Among Urban Poor Children Under Five in Kuala Lumpur, Malaysia: A Two-armed Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a Positive Deviance Program in Reducing Childhood Undernutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Gan Wan Ying, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JKEUPM-2020-349
Record Dates: First submitted 2020-12-20; First posted 2020-12-30 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition, Child
Keywords: Child undernutrition; Positive deviance; Urban poor children; Stunting; Wasting; Weight gain
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders; Cachexia; Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group refers to mother-child dyads who will be participating in a nutrition program consisting of nutrition education and cooking sessions for 3 months.
  Interventions: Behavioral: Nutrition program developed using positive deviance approach
- Comparison group (No Intervention): The comparison group will not receive any intervention but will be provided with the developed educational materials used in the program after the program has been completed.

INTERVENTIONS:
Behavioral: Nutrition program developed using positive deviance approach — It is a 3-month nutrition program including nutrition education session and rehabilitation session. The education session consists of half hour education lesson and one and half hours peer-led cooking session. The cooking demonstration will be led by volunteers from PD family. Participating mothers will need to bring along their children during this session, prepare meal according to pre-planned menu and feed their children with the prepared meal after cooking as snack or additional meal. The rehabilitation session will be the rest of the days following each education session until the next education session. Growth monitoring session will also be conducted in each session, whereby mothers will be taught and trained to weigh their children.
  Arms: Intervention group

SUMMARY:
Globally, childhood malnutrition remains a public health concern. Malnutrition can be diverse from undernutrition to overnutrition. A young child, primarily refers to those under the age of 5, is suffering from undernutrition when the child is lacking of adequate nutrition that necessary for proper growth and health due to direct or indirect causes such as not having enough food. In fully urbanized area such as Kuala Lumpur, urban poor children tend to face greater deprivations such as lower education and poor health which significantly influence their daily diet and nutritional status. Hence, urban poor children who are living and growing up in such underprivileged environment should not be neglected. Since young children are generally depending on maternal feeding for daily diet, intervention that focus on encouraging positive change in maternal feeding practices might be efficient in reducing childhood undernutrition. The positive deviance (PD) approach may consider as a better alternative to empower mothers by promoting new behaviour to feed their children. Hence, this study aims to evaluate the effectiveness of a nutrition program using PD approach in reducing undernutrition among urban poor children aged 3 to 5 years old in Kuala Lumpur.

DETAILED DESCRIPTION:
Background:

Undernourished children who fail to grow in height and weight as other normal children can be underweight, stunting or wasting. In fully urbanized area such as Kuala Lumpur in Malaysia, the consequences of undernutrition are more detrimental in urban poor young children. Since young children are generally depending on maternal feeding for daily diet, alternative intervention that focus on encouraging positive change in maternal behaviour when feeding children might be efficient in reducing childhood undernutrition. The positive deviance (PD) approach is one such alternative intervention. This approach emphases the identification of positive deviant, individuals who successfully discover a way to solve a problem by performing some uncommon but advantageous actions or behaviours in the same underprivileged environment as their peers. In the context of child nutrition, positive deviance is more frequently referred to as adaptive child care practices, positive hygiene practices and feeding practices that enable children to develop appropriately in a harsh environment with limited resources. The nutrition program developed using this approach helps to discover positive deviant, spread local wisdom from mothers of well-nourished children to mothers of undernourished children, and initiate positive behavioural change as a preliminary step to promote healthy weight gain in children.

Methods:

This is a mixed method study which will be carried out in two phases. Phase I of the study will involve focus group discussion (FGD) with semi-structured interview to explore maternal feeding practices and also foods being fed to children. Mothers of children aged 3 to 5 years old will be recruited through purposive sampling or until saturation point is reached. Phase II of the study will involve a two-armed randomized controlled trial to evaluate effectiveness of nutrition program. A total of 164 mother-child dyads will be recruited, in which 82 of them will be recruited separately and randomly from different PPR flats with 1:1 allocation to form intervention and comparison groups. Ethical approval will be obtained from the Ethics Committee for Research Involving Human Subjects Universiti Putra Malaysia (JKEUPM). Permission to conduct this study in PPR flats and the list of PPR flats in KL will be obtained from the Kuala Lumpur City Hall. Intervention group will need to participate in a nutrition program for 3 months that consists of education session with peer-led cooking session and rehabilitation session. The comparison group will be given all the materials used in the program for reference after the last data collection. The height and weight of children will be measured by researcher. Mothers will be interviewed on the dietary intake of their children. Mothers will also need to answer a Malay language self-administered questionnaire to obtain information on socio-demographic characteristics, nutrition knowledge and food security status. These measurements will be taken at the baseline (before intervention), immediate post-intervention and 3-month post-intervention for both intervention and comparison groups.

ELIGIBILITY:
For Phase 1:

Inclusion Criteria:

* Malaysian
* Children aged 3 to 5 years old
* Mothers aged above 18 years old
* Living in public low-cost PPR flat

Exclusion Criteria:

* Children who are taken care by other adults rather than mothers such as father, grandparents and caregivers
* Mothers with mental disabilities
* Children with history of chronic diseases including congenital heart disease, liver disease, renal failure or sickle cell disease and any congenital abnormalities
* Children who are under treatment for communicable disease such as measles and chickenpox
* Children with learning disabilities
* Mother-child dyads involved in any other intervention or clinical research
* Children who are overweight or obese

The respondents' selection criteria in Phase 2 are almost similar as in Phase 1 except for the second inclusion criterion that is related to children. In Phase 2, only undernourished children (either underweight, stunting or wasting) aged 3 to 5 years old will be recruited in order to evaluate the effectiveness of the intervention in this particular group. The exclusion criteria in Phase 2 are similar to the exclusion criteria in Phase 1.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in body weight after 3 months of intervention in children | 3 months
  body weight in kg
Changes in weight-for-age z score after 3 months of intervention in children | 3 months
  weight-for-age z score in standard deviation
Changes in height-for-age z score after 3 months of intervention in children | 3 months
  height-for-age z score in standard deviation
Changes in weight-for-height z score after 3 months of intervention in children | 3 months
  weight-for-height z score in standard deviation
Changes in dietary intake after 3 months of intervention in children | 3 months
  24-hour diet recall (3 days) in kcal
Changes in diet quality after 3 months of intervention in children | 3 months
  Healthy Eating Index (HEI) for Malaysians; composite HEI scores range from 0 to 100%; score <51% indicates poor diet quality, 51 to 80% indicates diet required improvement, and >80% indicates good diet quality

SECONDARY OUTCOMES:
Changes in nutrition knowledge after 3 months of intervention in mothers | 3 months
  20-item nutrition knowledge questionnaire; total scores range from 0 to 20 marks; higher score indicates good knowledge
Assessment of food security level after 3 months of intervention in mothers | 3 months
  6-item USDA Short Form Food Security Survey Module; It consists of affirmative responses such as 'always', 'sometimes', and 'yes', as well as non-affirmative responses such as 'never', 'no', and 'don't know'. An affirmative response is given a score of 1 and a non-affirmative response is given a 0 score. The possible total scores range from 0 to 6, and a score of 2 or higher indicates food insecurity

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ying Gan, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- PPR, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albanna, B., & Heeks, R. (2019). Positive deviance, big data, and development: A systematic literature review. Electronic Journal of Information Systems in Developing Countries, 85(1), e12063. https://doi.org/10.1002/isd2.12063
- [Background] Herington, M. J., & Fliert, E. Van De. (2017). Positive deviance in theory and practice : A conceptual review. Deviant Behavior, 39(5), 664-678. https://doi.org/10.1080/01639625.2017.1286194
- [Background] Schooley J, Morales L. Learning from the community to improve maternal-child health and nutrition: the Positive Deviance/Hearth approach. J Midwifery Womens Health. 2007 Jul-Aug;52(4):376-83. doi: 10.1016/j.jmwh.2007.03.001. PMID 17603960
- [Background] Sternin, M., Sternin, J., & Marsh, D. (1998). Designing a community-based nutrition program using the hearth model and the positive deviance approach - A field guide. Save the Children Federation.
- [Background] The CORE group. (2002). Positive deviance / Hearth essential elements: A resource guide for sustainably rehabilitating malnourished children. CORE group.
- [Derived] Chek LP, Gan WY, Chin YS, Sulaiman N. A nutrition programme using positive deviance approach to reduce undernutrition among urban poor children under-five in Malaysia: A cluster randomised controlled trial protocol. PLoS One. 2022 Oct 13;17(10):e0275357. doi: 10.1371/journal.pone.0275357. eCollection 2022. PMID 36227928